CLINICAL TRIAL: NCT01079221
Title: Effects of Knee-extensor Exercise Training in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 42009297
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2016-08-02 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: exercise; Knee extensor
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Knee extensor exercise training (Experimental): High intensity aerobic knee-extensor exercise training
  Interventions: Behavioral: High intensity knee-extensor training

INTERVENTIONS:
Behavioral: High intensity knee-extensor training — High intensity aerobic knee-extensor exercise training, 4x 3 minutes interval training at < 90 % of peak power, 3 days/week for 6 weeks

SUMMARY:
COPD patients have a reduced exercise tolerance due to a ventilatory limitation.

Several studies have shown altered skeletal muscle function. The investigator will study the physiological response to knee-extensor exercise in COPD patients.

DETAILED DESCRIPTION:
Reduced exercise tolerance is one of the hallmarks of COPD. The principal causes for exercise intolerance are ventilatory limitation leading to deconditioning and inactivity. However the weak correlation between exercise capacity and FEV1 implies that other factors than reduced pulmonary function contribute to this impairment as well. Several studies have found changes in skeletal muscle, with fibre shift, increased oxidative stress, increased inflammatory cytokines and impaired mitochondrial function, suggesting a lower limb dysfunction.

Numerous exercise studies in COPD patients have shown physiological and physiological benefits of training and endurance training is now regarded as an important part in pulmonary rehabilitation.

In this study we investigate training effects in patients with moderate to severe COPD with special focus on skeletal muscle.

COPD patients will perform high intensity aerobic interval knee-extensor exercise training 3 days/week for six weeks . At baseline and follow-up, muscle oxygen consumption and mitochondrial respiration will be measured.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis with FEV1<70% exp, FEV1%FVC <70 %
* Age> 50 years

Exclusion Criteria:

* Heart failure
* Symptomatic coronary artery disease
* Cancer
* Alcohol and drug abuse
* Severe mental illness
* Lower respiratory illness
* Participation in exercise- or lung rehabilitation program last 3 months
* pregnancy
* oral steroid use

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Peak power | At inclusion and after 6 weeks of training

SECONDARY OUTCOMES:
Mitochondrial respiration, Vmax | At inclusion and after 6 weeks of training

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, PhD prof., Study Director — Norwegian University of Science and Technology

REFERENCES:
- [Result] Bronstad E, Rognmo O, Tjonna AE, Dedichen HH, Kirkeby-Garstad I, Haberg AK, Ingul CB, Wisloff U, Steinshamn S. High-intensity knee extensor training restores skeletal muscle function in COPD patients. Eur Respir J. 2012 Nov;40(5):1130-6. doi: 10.1183/09031936.00193411. Epub 2012 Mar 9. PMID 22408206